CLINICAL TRIAL: NCT01319968
Title: Postpartum Dyspareunia Resulting From Vaginal Atrophy: Prevalence, Characteristics and Risk Factors
Brief Title: Postpartum Dyspareunia Resulting From Vaginal Atrophy
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MMC11030-2011kCTIL
Record Dates: First submitted 2011-03-20; First posted 2011-03-22 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2012-04

CONDITIONS: Vulvovaginal Atrophy; Dyspareunia Among Puerperal Women
Keywords: Postpartum dyspareunia; Vaginal atrophy
MeSH Terms: interventions — Estriol; Vaginal Creams, Foams, and Jellies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Vaginal smears for cytology and pH measurment.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Postpartum patients: 100 postpartum women attending the clinic for their postpartum visit will be evaluated for vaginal atrophy, vaginal symptoms and dyspareunia.
  Interventions: Drug: Estriol 0.1% vaginal cream

INTERVENTIONS:
Drug: Estriol 0.1% vaginal cream — Patients with both vulvovaginal atrophy (according to cytologic criteria) and dyspareunia will apply 0.5 ml of the cream (0.5 mg) to the vulvar vestibule once daily for one month and will return for check-up visit. In case both atrophy and dyspareunia will resolve, treatment with the cream will be continued 3 times a week.
  Other Names: Ovestin vaginal cream

SUMMARY:
Postpartum dyspareunia (PD) is a recognized phenomenon: it is estimated that 50-60% of women have dyspareunia 6 to 7 weeks following delivery, and 33% and 17% will still report pain during intercourse three and six months after delivery, respectively.

Studies that evaluated the prevalence and the causes for PD referred primarily to obstetric trauma, such as vaginal tears, episiotomy, the mode of repair and damage to the pelvic floor muscles as probable causes for PD. These studies did not refer to estrogen deficiency and the possible effect of breastfeeding on vaginal atrophy and its contribution to PD. Comparison between vaginal deliveries and cesarean sections revealed that there is no difference in the prevalence of PD between the two groups, and according to these findings it can be assumed that the mechanical trauma to the vagina and pelvic floor during delivery is not the main cause for the development of PD.

Vaginal atrophy due to estrogen deficiency is a common cause for postmenopausal dyspareunia. With estrogen deficiency, profound changes occur in the vagina: vaginal mucosa becomes thin and pale or hyperemic and loose her flexibility. Blood flow decreases, normal vaginal discharge is reduced, and maturation of epithelial cells do not take place in the absence of estrogen. Women with estrogen deficiency may complain of dryness, pruritus, irritation, burning, dysuria, pain and dyspareunia. These changes are reversible by estrogen, given systemically or topically, and cause resolution of clinical findings, as well as disappearance of symptoms in several weeks.

Similar to postmenopausal patients, breastfeeding women immediately after delivery, experience decline of estrogen levels, and this decline may persist as long as lactation is continued. Therefore, many women after delivery may experience vaginal atrophy due to transitional lack of estrogen. It is possible that this atrophy is the cause for the high rate of PD.

Our clinical experience shows that many women present with postpartum dyspareunia with vaginal atrophy, and that vaginal atrophy is responsible for part or most of their complaints. Although most gynecologists recognize atrophy easily in menopausal women, vaginal atrophy is not recognized correctly in most puerperal patients and therefore do not receive attention and proper treatment.

The aim of the study is to characterize the phenomenon of postpartum vaginal atrophy in terms of prevalence, risk factors and duration, and the association between vaginal atrophy and postpartum dyspareunia.

We also intend to evaluate the effect of vaginal treatment with estriol cream 0.1% (Ovestin cream) on postpartum dyspareunia.

The study will expand our knowledge regarding postpartum dyspareunia and will enable formulating recommendations for evaluation and treatment of PD.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, puerperal women who will be willing to participate, over 18 years old.

Exclusion Criteria:

* Patients with puerperal complications such as: bleeding, fever, endometritis.
* Patients with significant systemic diseases.
* Patients who conceive again during the study.
* Patients who are not willing to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 postpartum women attending the clinic for their postpartum visit
Sampling Method: Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2011-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Prevalence of vulvovaginal atrophy among puerperal women | one year
  Prevalence of vulvovaginal atrophy due to estrogen deficiency among puerperal women, according to cytological parameters.

SECONDARY OUTCOMES:
Prevalence of dyspareunia among women with puerperal vaginal atrophy. | one year
  Prevalence and cause of dyspareunia among puerperal women with and without vaginal atrophy will be assesed
Effect of treatment with topical estrogen on dyspareunia. | 2 months from begining of treatment
  The effect of vaginal estrogen cream on the prevalence of atrophy, its effect on postpartum dyspareunia and side effects.

CONTACTS AND LOCATIONS:
Overall Officials: Ahinoam Lev-Sagie, MD, Principal Investigator — Clalit Health Services
Locations (2):
- Israel (2):
  - Clalit Women's Health Center, Jerusalem
  - Clalit Women's Health Center, Modiin

REFERENCES:
- [Background] Wisniewski PM, Wilkinson EJ. Postpartum vaginal atrophy. Am J Obstet Gynecol. 1991 Oct;165(4 Pt 2):1249-54. doi: 10.1016/s0002-9378(12)90737-1. PMID 1659199
- [Background] Signorello LB, Harlow BL, Chekos AK, Repke JT. Postpartum sexual functioning and its relationship to perineal trauma: a retrospective cohort study of primiparous women. Am J Obstet Gynecol. 2001 Apr;184(5):881-8; discussion 888-90. doi: 10.1067/mob.2001.113855. PMID 11303195
- [Background] Carroli G, Mignini L. Episiotomy for vaginal birth. Cochrane Database Syst Rev. 2009 Jan 21;(1):CD000081. doi: 10.1002/14651858.CD000081.pub2. PMID 19160176